CLINICAL TRIAL: NCT03442647
Title: Dynamic Measurement of Renal Functional Reserve as a Predictor of Long-Term Renal Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Mueller (Other)
Responsible Party: Sponsor-Investigator, Thomas Mueller, Prof. Dr., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-01839
Record Dates: First submitted 2018-02-05; First posted 2018-02-22 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Adult Polycystic Kidney Disease; Kidney Neoplasms; Kidney Dysfunction
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Kidney Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Living donors (Active Comparator): sinistrin clearance dynamic measurement
  Interventions: Diagnostic Test: sinistrin clearance dynamic measurement
- ADPKD patients (Active Comparator): sinistrin clearance dynamic measurement
  Interventions: Diagnostic Test: sinistrin clearance dynamic measurement
- Patients with primary renal tumor (Active Comparator): sinistrin clearance dynamic measurement
  Interventions: Diagnostic Test: sinistrin clearance dynamic measurement

INTERVENTIONS:
Diagnostic Test: sinistrin clearance dynamic measurement — sinistrin clearance measurements will be performed before and 90 min after oral protein load

SUMMARY:
The number of people with kidney disease is constantly rising and renal failure represents one of the major health care burdens globally. An accurate measurement of kidney function is urgently needed to better understand and treat loss of renal function. Kidneys have an intrinsic reserve capacity to respond to a higher work load by increasing filtration in their nephrons. The number of nephrons and their reserve capacity define how well kidneys can adapt to an increased demand and disease.

The degree of renal reserve capacity becomes particularly important when the number of functioning nephrons is significantly reduced either due to surgical removal of one kidney as in living kidney donation or in tumor nephrectomy or due to progressive injury as in autosomal dominant polycystic kidney disease (ADPKD). A reduced functional reserve likely reflects an impaired adaptive capacity and increased risk of accelerated loss of function in the remaining single kidney or in kidneys exposed to a disease. Despite the importance of accurately measuring baseline and reserve capacity renal function, due to the time- and laborintensive procedure, in clinical routine this testing is rarely done.

Investigators aim to measure renal functional reserve (RFR) and loss of function in patients undergoing nephrectomy (living kidney donors and renal tumor patients) as well as in patients with ADPKD.

The results should provide evidence whether renal functional reserve indeed predicts adaptive capacity and functional loss after removal of a healthy kidney (living donors), of a tumor kidney (cancer patients) or in progressive kidney disorders (ADPKD patients).

Investigators are confident that the proposed project will enhance the understanding of progressive kidney disease and with this improve donor safety, planning of tumor nephrectomy, and prediction of renal functional loss as well as provide a strong argument that dynamic renal function testing, i.e. accurate measurement of baseline and reserve capacity, is necessary in certain disease entities.

DETAILED DESCRIPTION:
The measurement of RFR will be performed by dynamic testing of the changes in baseline glomerular filtration rate (GFR) induced by an oral protein load. Sinistrin (a polyfructosan with identical clearance characteristics to inulin) will be used to measure GFR.

ELIGIBILITY:
Inclusion Criteria:

* Potential living kidney donor
* Patients with diagnosed ADPKD
* Patients with primary kidney tumor requiring nephrectomy
* Female and male patients over 18 years of age

Exclusion Criteria:

* Bilateral kidney tumor
* Kidney metastases of a tumor of other origin
* Renal failure that requires dialysis
* Pregnant patient
* Incomplete medical records
* Patients with diabetes mellitus
* Patients who cannot tolerate iv fluids
* Hypersensitivity to the active substance (sinistrin) or to any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2018-08-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
RFR predicts renal functional decline | up to 8 months
  Sinistrin levels in plasma before and after oral protein load. Participants with impaired RFR are expected to have higher sinitrin levels in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Mueller, Prof., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland